CLINICAL TRIAL: NCT02699463
Title: Assessment of the Effect of Positive Airway Pressure on Energy and Vitality in Mild Obstructive Sleep Apnea Patients: The Merge Study
Brief Title: Assessment of the Effect of PAP on Energy and Vitality in Mild OSA Patients: The Merge Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA200216
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continous Positive Airway Pressure (Active Comparator): Participants in this group will use CPAP therapy, nightly, for the 3 month duration of the trial
  Interventions: Device: Continous Positive Airway Pressure
- Control Group (Placebo Comparator): Participants will receive standard care (Sleep hygiene counseling) during the study.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Continous Positive Airway Pressure — CPAP refers to the application of positive airway pressure through a mask and tubing to splint a patients throat open at night. CPAP is considered standard treatment for OSA
  Other Names: CPAP
  Arms: Continous Positive Airway Pressure
Other: Control Group — Standard sleep hygiene counseling as per published guidelines
  Arms: Control Group

SUMMARY:
The investigators wish to prospectively determine the response to CPAP in patients presenting with mild OSA. In many healthcare systems, patients with mild OSA (AHI 5-15) are not reimbursed for treatment. Although some evidence exists of the benefits of treating mild OSA when scoring as per AASM 2007 criteria, more evidence is needed. The investigators wish to add to this pool of knowledge and also increase the inclusion criteria to include the AASM 2012 definition of mild OSA. By including the 2012 AASM definition of mild OSA, the investigators will add novel information to the field by assessing the benefits of treatment in both sub-groups of mild OSA.

DETAILED DESCRIPTION:
Patients who visit their local sleep service for OSA investigation, and are found to have mild OSA (AHI ≤ 15) from an Apnealink polygraphy (PG) home sleep test, scored as per AASM 2007 and/or AASM 2012, will be invited to take part in the study (pre-screening).

At the study visit, informed consent, baseline demographics, and standardised questionnaires will be administered. Participants will then be randomised to a CPAP treatment group or control group.

After 3 months, participants will be asked to repeat the standardised questionnaires, the trial will then be complete and they will return to routine clinical care.

ELIGIBILITY:
Study Inclusion Criteria

* Aged ≥ 18 and ≤ 80
* Ability and willingness to provide written informed consent
* AHI ≤ 15 as per AASM 2007 scoring criteria
* Ability to tolerate a CPAP one hour long run in test

Exclusion Criteria:

* The presence of unstable cardiac disease
* Inability to give fully informed consent
* Supplemental oxygen
* Secondary sleep pathology e.g. Periodic Limb Movement Syndrome, Narcolepsy, Circadian Disorder, obesity hypoventilation syndrome
* ESS ≥ 15, or concerns about sleepy driving from physician/ sleep lab staff
* BMI ≥ 40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2016-12; Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Morrell, Prof, Principal Investigator — Imperial College London
Locations (11):
- United Kingdom (11):
  - Freeman Hospital, Newcastle upon Tyne, Newcastle
  - Blackpool Teaching Hospital, Blackpool
  - Papworth Hospital, Cambridge
  - Tayside Health Board, Ninewells Hospital, Dundee
  - Aintree University Hospital, Liverpool
  - Royal Brompton Hospital, Imperial College London, London
  - Guys & St Thomas Hospital, London
  - Oxford Centre for Respiratory Medicine, Oxford
  - Derriford Hospital, Plymouth
  - Lister Hospital, Stevenage
  - Taunton and Somerset Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wimms AJ, Kelly JL, Turnbull CD, McMillan A, Craig SE, O'Reilly JF, Nickol AH, Hedley EL, Decker MD, Willes LA, Calverley PMA, Benjafield AV, Stradling JR, Morrell MJ; MERGE trial investigators. Continuous positive airway pressure versus standard care for the treatment of people with mild obstructive sleep apnoea (MERGE): a multicentre, randomised controlled trial. Lancet Respir Med. 2020 Apr;8(4):349-358. doi: 10.1016/S2213-2600(19)30402-3. Epub 2019 Dec 2. PMID 31806413

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 301 participants were randomised. 233 patients formed the primary analysis group. Of those, 115 were allocated to the CPAP group and 118 were allocated to standard care. The remaining 68 patients were not analysed as part of the primary analysis but were analysed for secondary analysis.
Period: Overall Study
Arm/Group | Continous Positive Airway Pressure | Control Group
Started | 115 | 118
Completed | 100 | 109
Not Completed | 15 | 9
Not completed — Lost to Follow-up | 11 | 8
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continous Positive Airway Pressure | Control Group | Total
Number analyzed (Participants) | 115 | 118 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (11.3) | 50.2 (12.1) | 50.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 37 | 71
  Male | 81 | 81 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 105 | 103 | 208
  non-white | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Using the Energy and Vitality Subscale of the Short Form 36 (SF-36) Questionnaire
Description: The Short Form 36 (SF-36) questionnaire measures quality of life through a range of questions asking about patients physical and mental functioning. Specifically, the Energy and Vitality subscale records patients perceptions of their levels of energy and fatigue. Participants were administered the Short Form 36 (SF-36) questionnaire at baseline and 3 months. The change in score (value at 3 months minus value at baseline) was compared between the CPAP group and the Control group.
  In the SF-36 Energy and Vitality subscale, an increase in score indicates improvement, with a minimum score of 0 and a maximum score of 100 possible.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Continous Positive Airway Pressure | Control Group
Number analyzed (Participants) | 115 | 118
score on a scale | 7.5 [6.0 to 9.0] | 0 [-1.5 to 1.5]
Statistical Analysis 1: Comparison: Continous Positive Airway Pressure vs Control Group; Test type: Superiority; p < 0.01, ANCOVA — The calculated p-value was <0.01

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Continous Positive Airway Pressure | Control Group
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/118
Serious Adverse Events (participants affected / at risk) | 1/115 | 2/118
Other Adverse Events (participants affected / at risk) | 9/115 | 13/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continous Positive Airway Pressure (N=115) | Control Group (N=118)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
hospitalization for dizziness, existing cardiac condition (Cardiac disorders) | 0 (0) | 1 (1)
symptoms of transient ischemic attack (TIA) (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continous Positive Airway Pressure (N=115) | Control Group (N=118)
dizziness (Cardiac disorders) | 3 (4) | 0 (0)
exacerbation of pre-existing condition (General disorders) | 2 (2) | 8 (8)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
physical accident (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
virus (Infections and infestations) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT02699463/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT02699463/SAP_001.pdf